CLINICAL TRIAL: NCT04251351
Title: Evaluating the Renoprotective Effect of Paracetamol in Paediatric Severe Malaria: a Randomised Controlled Trial
Brief Title: Effect of Paracetamol on Kidney Function in Severe Malaria
Acronym: PROTECtS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other); Kinshasa Medical Oxford Research Unit (Unknown)
Responsible Party: Principal Investigator, Katherine Plewes, MD PhD, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H19-03570
Record Dates: First submitted 2019-12-17; First posted 2020-01-31 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Severe Malaria; Malaria,Falciparum; Acute Kidney Injury; Paracetamol
Keywords: Severe Malaria; Falciparum; Paracetamol; Renoprotection; Acute Kidney Injury
MeSH Terms: conditions — Malaria; Malaria, Falciparum; Acute Kidney Injury | interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: Prior to randomization, participants will be stratified into two groups: (i) Patients with no acute kidney injury (AKI) at enrolment, and (ii) Patients with AKI at enrolment. Both groups will be randomised into two arms:
  Arm 1: Paracetamol 15 mg/kg/dose 6 hourly for 72 hours
  Arm 2: Mechanical antipyresis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Paracetamol 15 mg/kg/dose 6 hourly for 72 hours
  Interventions: Drug: Paracetamol
- Arm 2 (Sham Comparator): Mechanical antipyresis (i.e. loose clothing, tepid sponging, fanning and cooling blanket) if fever in the first 72 hours.
  Interventions: Procedure: Mechanical antipyresis

INTERVENTIONS:
Drug: Paracetamol — Paracetamol 15 mg/kg/dose IV 6 hourly for 72 hours
  Other Names: Acetyl-Para-Aminophenol (APAP); Acetaminophen
  Arms: Arm 1
Procedure: Mechanical antipyresis — Mechanical antipyresis (i.e. loose clothing, tepid sponging, fanning and cooling blanket) if fever in the first 72 hours.
  If a temperature >38.5°C persists despite mechanical antipyresis, or if deemed necessary by the treating clinician, then paracetamol can be administered according to local practice (paracetamol IV 15 mg/kg as needed).
  Arms: Arm 2

SUMMARY:
A randomised open labeled, parallel-group, controlled trial to assess the efficacy of paracetamol to reduce kidney dysfunction caused by cell-free haemoglobin-mediated oxidative damage in paediatric patients with falciparum malaria complicated by intravascular haemolysis.

DETAILED DESCRIPTION:
Kidney dysfunction is an independent predictor of mortality in both adults and children with severe malaria. In the largest studies of paediatric severe malaria, approximately 25% of children had kidney dysfunction and these patients accounted for roughly 50% of total deaths.

Although the multifactorial mechanism of severe malaria-associated AKI has primarily been studied in adults, evidence suggests that similar mechanisms of renal injury are involved in paediatric severe malaria. Cell-free haemoglobin (CFH) -mediated oxidative damage has recently been recognized as an important pathway in a range of common conditions, including rhabdomyolysis, primary pulmonary graft dysfunction, and haemolytic disorders, such as post-cardiac surgery, and malaria. During malaria infection, there is haemolysis of parasitized and uninfected red blood cells (RBCs). CFH-mediated lipid peroxidation generates F2-isoprostanes (F2-IsoPs) and isofurans (IsoFs), which are considered robust in vivo measures of oxidative stress. F2-IsoPs are potent renal vasoconstrictors that act via thromboxane A2 receptors. Both F2-IsoPs and IsoFs have been associated with AKI in patients with rhabdomyolysis, sepsis, adults with severe malaria and haemolysis post-cardiopulmonary bypass (CPB). Further, elevated haemin and CFH concentrations were associated with mortality. In a cohort of children with severe malaria, elevated haem-to-haemopexin ratio was associated with stage 3 AKI, and 6-month mortality. These studies demonstrate that intravascular haemolysis occurs with increasing severity in paediatric malaria. Haem redox cycling between ferric (Fe3+) and ferryl (Fe4+) states generates globin radicals, inducing lipid peroxidation. These data suggested that haemolysis induces oxidative damage, and CFH-mediated oxidative damage contributes to AKI complicating paediatric malaria.

A novel mechanism of paracetamol was recently demonstrated, showing that paracetamol acts as a potent inhibitor of haemoprotein-catalyzed lipid peroxidation, by reducing ferryl haem to its less toxic ferric state and quenching globin radicals. We hypothesize that this novel inhibitory mechanism of paracetamol may provide renal protection in children with severe malaria by reducing the haemoprotein-induced lipid peroxidation. As there is currently no consensus that exists concerning adequate medical treatment for severe malaria complicated by intravascular haemolysis and AKI, the potential application of this safe and extensively used drug would be of great benefit.

The study will be a randomised, open-labelled, controlled trial. Randomisation will be stratified into two groups : (i) Patients with no acute kidney injury (AKI) at enrolment, and (ii) Patients with AKI at enrolment. Both groups will be randomised into two arms: Arm 1: Paracetamol 15 mg/kg/dose 6 hourly for 72 hours Arm 2: Mechanical antipyresis if fever in the first 72 hours. All patients will receive intravenous artesunate followed by artemether-lumefantrine as soon as they are able to take oral medication or according to medical judgment.

The study will be conducted at the Kinshasa Medical Oxford Research Unit (KIMORU, Democratic Republic of the Congo, DRC). The recruitment phase of the study is expected to last 18 months, from September 2021 - February 2022. The total time to complete the study will be approximately 3 years.

Funder: Canadian Institutes of Health Research

CIHR grant reference number : PJT-162116

UBC grant number: 20R01487

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, patients aged 1 to ≤ 14 years
2. Severe P. falciparum malaria, confirmed by positive blood smear with asexual forms of P. falciparum or positive PfHRP2 rapid diagnostic test (RDT).

   Pre-specified modified criteria for severe falciparum malaria

   Upon hospital admission, asexual parasitaemia plus at least ONE of the following:
   * Glasgow coma score < 11/15 or Blantyre coma score <3/5 in pre-verbal children
   * Generalized convulsions (≥2 in 24 hours)
   * Jaundice (visible jaundice)
   * Severe anaemia (HCT <15%/Hb<5 g/dL: aged <12) Severe anaemia (HCT <20%/Hb<7 g/dL: aged ≥12)
   * Hyperparasitaemia (>10%)
   * Hypoglycaemia (glucose < 2.2 mmol/L; <40 mg/dL)
   * Kidney dysfunction (blood urea > 20 mmol/L)
   * Acidosis (venous bicarbonate <15 mmol/L or base excess less than -3.3mEq/L)
   * Venous lactate > 5 mmol/L
   * Shock (systolic blood pressure < 70 mmHg (<12 years) <80 mmHg (≥12 years) with cool extremities or capillary refill >3 seconds)
   * Respiratory distress (costal indrawing, use of accessory muscles, nasal flaring, deep breathing or severe tachypnea (respiratory rate>ULN for age)
   * Spontaneous bleeding
   * Prostration (inability to set upright, or drink)* Abbreviations: HCT, haematocrit; Hb, haemoglobin; *cannot be only severity criteria
3. Temperature >38°C on admission or fever during the preceding 48 hours.
4. Less than 24 hours of antimalarial therapy
5. Attending caregiver of participant willing and able to give informed consent for participation in the study

Exclusion Criteria:

The participant may not enter the trial if ANY of the following apply:

1. Contraindication or known allergy to paracetamol
2. Known chronic liver disease or tender hepatomegaly
3. Known chronic kidney disease, history of renal replacement therapy or renal biopsy
4. Participants who are already enrolled in another research trial involving an investigational product or have participated to the same study before

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 460 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Acute kidney injury (AKI) or death among patients enrolled without AKI (Composite outcome) | during first 7 days of enrolment
  Composite outcome of development of AKI (defined as creatinine ≥26.5 µmol/L or ≥1.5x baseline), or death at any timepoint
Acute kidney injury (AKI) progression or death among patients enrolled with AKI (Composite outcome) | during first 7 days of enrolment
  Composite outcome of worsening of AKI (defined as creatinine ≥2x baseline, or ≥3x baseline, or initiation of RRT or eGFR <35 ml/min/ 1.73 m2) or death at any timepoint.

SECONDARY OUTCOMES:
Number of patients with serious adverse events | AST/ALT/total bilirubin during the first 5 days from enrolment; mortality assessed Day 0 to 7.
  Number of patients with serious adverse events (mortality and/or hepatotoxicity, as defined by Hy's Law).
Proportion of patients who develop Major Adverse Kidney Events (MAKE) composite | 90 days
  Major Adverse Kidney Events (MAKE) composite, defined as ≥ 1 efficacy renal endpoints: (i) death, (ii) need for renal replacement therapy, (iii)≥ 50% reduction in eGFR from baseline to 90 days.
Fever clearance time | 6-hourly temperature assessments during first 7 days from enrolment
  Time taken for aural temperature: (i) to fall < 37.5°C (FCT-A), and (ii) to fall < 37.5°C and remain there for >24 h (FCT-B)
Coma recovery | 6-hourly GCS/BCS assessments during first 7 days from enrolment
  Time until Glasgow Coma Score (GCS) return to 15 (or Blantyre Coma Score (BCS) return to 5 in preverbal children)
Longitudinal change in renal function | During the first 7 days from enrolment
  As measured by creatinine concentration (umol/L)
Longitudinal change in markers of hemolysis | during the first 3 days from enrolment
  As measured by cell-free haemoglobin (ug/mL), haemopexin (ug/mL), haptoglobin (ug/mL), haem (uM), F2-isoprostane (pg/mL) and isofurans (pg/mL) concentrations
Longitudinal change of endothelial activation | during the first 3 days from enrolment
  As measured by concentrations of angiopoietin-Tie2 pathway markers (i.e. Ang-1, Ang-2, sTie2, sTie1)
Longitudinal change of immune activation | during the first 3 days from enrolment
  As measured by soluble triggering receptor expressed on myeloid cells concentration (sTREM-1; pg/mL)
Longitudinal change of AKI biomarker | during the first 3 days from enrolment
  As measured by cystatin-C concentration (Cys-C; ug/mL)
Parasite (parasites/ul) clearance | 12-hourly parasitemia assessments during first 7 days from enrolment
  as measured by time until two consecutive negative smears (hours), and by rate using the parasite clearance estimator to determine slope half-life (hours) from 12-hourly parasite counts.
Exploratory analysis with sex | During first 7 days from enrolment
  Primary efficacy analyses will be analysed using a logistic regression model to obtain odds ratios, comparing the odds of a combined endpoint of kidney function deterioration or death between treatment groups. A multivariable model including an interaction term (sex and treatment) will be assessed in the primary analyses to explore potential differences between males and females.
Pharmacokinetic properties | during the first 24 hours from enrolment
  Population pharmacokinetic model (relative bioavailability, mean transit absorption time (hours), apparent oral elimination clearance (L/hours), apparent volume of distribution (L)
Pharmacokinetic properties | during the first 24 hours from enrolment
  Peak plasma concentration (Cmax; mg/L)
Pharmacokinetic properties | during the first 24 hours from enrolment
  Time to peak plasma concentration (Tmax; hours)
Pharmacokinetic properties | during the first 24 hours from enrolment
  Terminal elimination (t1/2; hours)
Pharmacokinetic properties | during the first 24 hours from enrolment
  Area under the plasma drug concentration-time curve (AUC0-24; mg×h×L-1)
Pharmacodynamic relationships | during first 7 days from enrolment
  Pharmacodynamic effects on creatinine concentration (mol/L)
Pharmacodynamic relationships | during first 7 days from enrolment
  Pharmacodynamic effects on liver toxicity, as measured by AST and ALT (U/L)
Pharmacodynamic relationships | during first 7 days from enrolment
  Pharmacodynamic effects on temperature (Celsius)
Pharmacodynamic relationships | during first 7 days from enrolment
  Pharmacodynamic effects on parasitemia, as measured by parasites/ul and slope half-life
Pharmacodynamic relationships | during first 7 days from enrolment
  Pharmacodynamic effects on GCS (or BCS in pre-verbal children)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Plewes, Dr., Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (1):
- The Kinshasa Medical Oxford Research Unit (KIMORU), Kinshasa, Congo, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Yes
Participant data and results from blood analyses stored in the database may be shared according to the terms defined in the MORU data sharing policy with other researchers to use in the future. Datasets will be de-identified to ensure patient privacy and confidentiality.
Time Frame: After completion of trial activities and reporting
Access Criteria: MORU Data Sharing Policy. (http://www.tropmedres.ac/data-sharing-policy)